CLINICAL TRIAL: NCT03492320
Title: Progression of Health Related Quality of Life of Patients Waiting for Total Knee Arthroplasty
Acronym: TKA HRQoL
Status: Completed | Type: Observational
Sponsor: Dr. Ho Ki Wai (Other)
Responsible Party: Sponsor-Investigator, Dr. Ho Ki Wai, Assistant Professor, Department of Orthopaedics & Traumatology; Director of MSc/PgD Programme in Musculoskeletal Medicine & Rehabilitation, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: CUHK_2013.381; CREC Ref. No. (Other: Joint CUHK-NTEC Clinical Research Ethics Committee)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Knee Arthroplasty; Knee Arthroplasty, Total; Knee Replacement, Total; Replacement, Total Knee; Total Knee Replacement; Health-Related Quality Of Life; Life Quality; Osteoarthritis Of Knee
Keywords: HRQoL; Quality of Life; End Stage Osteoarthritis; Total Knee Arthroplasty; WOMAC; SF 36; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health Quality of Life Questionnaire Assessment — Western Ontario and McMaster University Osteoarthritis Index (WOMAC), Self-Rated Questionnaire SF36 and Health Related Quality of Life (HRQoL) 15D questionnaire were used as outcome measurement for functionality and disability assessment.

SUMMARY:
To evaluate the progression on patients suffering from end stage OA whilst being on the waiting list for TKR

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) remains the surgical gold standard treatment for patients suffering from end stage osteoarthritis (OA) of the knee. However, due to the high demand and scarce medical resources, the waiting time for surgery is astoundingly lengthy. Controversies are shown on numerous studies on whether physical functionality and mental status decline or remain stable over the waiting period. This study aims to evaluate the progression on patients suffering from end stage OA whilst being on the waiting list for TKR.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with symptomatic osteoarthritis
2. Enlisted on the TKA surgical waiting list
3. Ethnic Chinese
4. Fluent in Cantonese

Exclusion Criteria:

1. Evidence of cognitive dysfunction like dementia
2. Surgery scheduled within 30 days
3. Severe co-morbidity preluding participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study aims to evaluate the progression on patients suffering from end stage OA whilst being on the waiting list for TKR. This was a prospective longitudinal study, involving patients with symptomatic osteoarthritis at Prince of Wales Hospital Hong Kong. This study was conducted from March 2013 to December 2016. By universal sampling, patients who had experienced symptomatic OA visiting the Li Ka Shing Orthopaedic Specialist out-patient clinic were screened by a research nurse or a research assistant based on the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | From March 2013 to December 2016
  Questionnaire
Self-Rated Questionnaire SF36 | From March 2013 to December 2016
  Questionnaire
Health Related Quality of Life (HRQoL) 15D | From March 2013 to December 2016
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ki Wai Ki Wai, Dr., Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided